CLINICAL TRIAL: NCT03679546
Title: EFFICACI : EFFicacy of Intravenous Infliximab Versus Vedolizumab After Failure of subCutaneous Anti-TNF in Patients With UlCerative Colitis : A Double Blinded Randomized Clinical Trial
Brief Title: EFFICACI : EFFicacy of Intravenous Infliximab Versus Vedolizumab After Failure of subCutaneous Anti-TNF in Patients With UlCerative Colitis
Acronym: EFFICACI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC17_8841_EFFICACI; 2018-002673-21 (EudraCT Number); 2018-66-PP (Other: CPP Sud-Est I)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; vedolizumab

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, double blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator will proceed to the patient randomization as follows :
  * The investigator fulfill the electronic case report form (eCRF)
  * The randomization will be performed through the eCRF.
  * A mail will be sent to the pharmacy that included the inclusion number of the patient, the group allocated and the dose of infliximab or vedolizumab to be infused.
  * A mail will be sent to the investigator that included only the inclusion number of the patient.
  The trial is conducted in a double-blind manner. The biostatistician who generated the randomization list, the person in charge of pharmacovigilance, the pharmacy of the clinical trials of the Rennes university hospital and the pharmacist of the recruiting center can have access to the arm of treatment under study.
  Patients and physicians will not know the nature of the molecules administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Infliximab : The treatment is infused at a dose of 5 mg/kg at week 0, 2 and 6 and then every 8 weeks.
  Interventions: Drug: Infliximab
- Vedolizumab (Experimental): Vedolizumab : The treatment is infused at a dose of 300 mg at week 0, 2 and 6 and then every 8 weeks.
  Interventions: Drug: Vedolizumab Injection

INTERVENTIONS:
Drug: Infliximab — Infliximab : The treatment is infused at a dose of 5 mg/kg at week 0, 2 and 6 and then every 8 weeks.
  Other Names: Infliximab injection
  Arms: Infliximab
Drug: Vedolizumab Injection — Vedolizumab : The treatment is infused at a dose of 300 mg at week 0, 2 and 6 and then every 8 weeks.
  Other Names: Vedolizumab
  Arms: Vedolizumab

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD) that results from immune dysregulation. Arguably, the development of Tumor Necrosis Factor (TNF) antagonists (including infliximab, adalimumab and golimumab) revolutionized the management of immune-mediated chronic diseases in the past two decades.

However, about one third of patients will not respond to a first anti-TNF treatment and 10% to 30% will loose response to anti-TNF during the follow-up.

Historically, a switch between anti-TNF was performed to recapture remission and response to anti-TNF. Recently, a new biologic therapy blocking another target has been approved and is now reimbursed during ulcerative colitis, namely vedolizumab. Vedolizumab is an anti-integrin agent avoiding the recruitment of lymphocytes specifically in inflamed gut tissue.

Emerging data suggest that a switch of therapeutic class (meaning a change of biologic target with Non-TNF-targeted biologic) in case of clinical failure or insufficient response to anti-TNF may be the best choice. This idea of a switch out of the anti-TNF class is also supported by data on drug monitoring that may help physician decision making in case of loss of response. However, no trial is currently available and ongoing to assess the best therapeutic strategy. The aim of the proposed study is to assess the best biological based strategy in patient losing response to a first subcutaneous anti-TNF (golimumab and/or adalimumab).

DETAILED DESCRIPTION:
Design :

A prospective, multicenter, randomized, double blind clinical trial

Primary objective :

To determine whether a non-TNF-targeted biologic (vedolizumab) is superior to infliximab to treat patient with UC losing response or with a primary failure to a first subcutaneous anti-TNF drug at week 14.

Secondary objective :

* To assess the rate of clinical response and remission at Week 54 in each group of treatments and the time to clinical response and remission from baseline ;
* To assess the changes in faecal calprotectin levels from baseline to week 14 and 54 according to treatment ;
* To assess the rate of colectomy and hospitalization in each treatment group ;
* To assess the rate of mucosal healing at week 14 and 54 in each group of treatments ;
* To assess the rate of loss of response in each group of treatments for patients responder after induction phase ;
* To assess the changes of quality of life indexes and the disability index from baseline to week 14 and 54 ;
* To determine the safety profile of each group of treatments ;
* To characterize the response in each group of treatments according to drug monitoring of the first anti-TNF agent ;
* To describe the pharmacokinetics of infliximab and vedolizumab as second-line treatment of UC and explore the sources of pharmacokinetic inter-individual variability ;
* To identify predictive factors of response to the treatment, including pharmacokinetic features

Expected findings and impact:

The patients include in the clinical will not lose any benefit since both treatments are actually indicated and effective in this condition. In both arm of treatment, patients will receive an effective treatment.

The study will optimize physician decision making to decrease the disease activity period in UC patients with known consequence such as hospitalisation, surgery, work cessations with related cost effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, non-lactating female;
* 18 years of age or older and less than 75 years ;
* Documented diagnosis of UC for at least 6 months ;
* Left side colitis or pancolitis ;
* Moderate to severe disease according to a Mayo score equal or above 6 with a Mayo endoscopic sub-score of 2 or 3 ;
* Active disease despite ongoing treatment with adalimumab or golimumab for at least 12 weeks (inadequate response, failure, loss of response or intolerance) ;
* Ability of the subject to participate fully in all aspects of this clinical trial ;
* Written informed consent must be obtained and documented ;
* Naïve to Janus kinase inhibitor (JAK inhibitor) ;
* Affiliation to the national health insurance.

Non inclusion Criteria:

* Contraindication to continue TNF antagonist (ongoing abscess(es), clinical suspicion of tuberculosis, past allergic reaction) ;
* Contraindication to vedolizumab treatment ;
* Steroid treatment > 20 mg/day for at least two weeks before baseline ;
* Proctitis ;
* Stoma ;
* Proctocolectomy or subtotal colectomy ;
* Planned surgery within the year of the trial ;
* Previous exposure to vedolizumab or infliximab ;
* History of cancer during the past 5 years ;
* Pregnancy or breastfeeding
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.
* Ongoing participation to another interventional study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Remission | Week 14
  The rate of patients with clinical and endoscopic steroid free-remission (Mayo score ≤ 2 without subscore > 1) at week 14

SECONDARY OUTCOMES:
Mayo score | Week 54
  Mayo score at week 54
Faecal calprotectin level | At week 14 and 54
  Faecal calprotectin level at week 14 and 54
Colectomy or hospitalization for disease flare | through study completion, an average of 1 year
  Colectomy or hospitalization for disease flare during the study period
Endoscopic subscore of the mayo Score | at week 14 and 54
  Endoscopic subscore of the mayo Score at week 14 and 54 Partial Mayo score at week 2, 6, 14, 54. Endoscopic subscore of the Mayo score : from 0 (better score) to 3 (worse score)
Partial Mayo score | at week 2, 6, 14, 54
  Partial Mayo score at week 2, 6, 14, 54. Partial Mayo score : from 0 (better score) to 9 (worse score)
Inflammatory Bowel Disease Questionnaire (IBDQ) index | at baseline week 14 and 54
  IBDQ index at baseline week 14 and 54
Inflammatory Bowel Disease-Disk (IBD-Disk) | at baseline week 14 and 54
  IBD-Disk at baseline week 14 and 54
Inflammatory Bowel Disease-Disability Index (IBD-DI) | at baseline week 14 and 54
  IBD-DI at baseline week 14 and 54
Adverse events | through study completion, an average of 1 year
  Rate and type of adverse events during the study period
Last trough concentration of the first subcutaneous agent | baseline
  Last trough concentration of the first subcutaneous agent at the time of the loss of response
anti-drug antibodies concentration | baseline
  anti-drug antibodies concentration at the time of the loss of response and
Blood trough concentration of infliximab or vedolizumab | at baseline, weeks 0, 2, 6, 14 and 54
  Trough concentration of infliximab or vedolizumab at each visit and anti-drug antibodies concentration (blood concentration)
Fecal trough concentration of infliximab or vedolizumab | at baseline, weeks 0, 2, 6, 14 and 54
  Trough concentration of infliximab or vedolizumab at each visit and anti-drug antibodies concentration (fecal concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOUGUEN, MD, Principal Investigator — Rennes University Hospital
Locations (19):
- France (19):
  - Centre Hospitalier Universitaire d'Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Assistance Publique des Hôpitaux de Paris - Hôpital Beaujon, Clichy
  - Assistance Publique des Hôpitaux de Paris - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Assistance Publique des Hôpitaux de Paris - Hôpital Saint-Louis, Paris
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No